CLINICAL TRIAL: NCT02050737
Title: Identification of Plasma Biomarkers in Early Detection of Colorectal Adenocarcinoma Recurrence (C-RAC Plasma Biomarker Study)
Brief Title: Plasma Biomarkers C-RAC, ICORG 12-27, V1
Status: Terminated | Type: Observational
Why Stopped: As per the HRBs new funding model, HRBs investment will not support costs associated with routine patient care or translational studies, biobanks, patient registries and questionnaires. Therefore, a decision was made to cease further study follow up.
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 12-27
Record Dates: First submitted 2014-01-23; First posted 2014-01-31 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: Curative resection; Adjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- A - due for adjuvant chemotherapy: Stage II/III colorectal cancer resectable disease due for adjuvant chemotherapy
- B - for observation only: Stage II colorectal cancer with resectable disease for observation only

SUMMARY:
This is an exploratory, translational, non-interventional and multi-centre clinical study.

DETAILED DESCRIPTION:
Cohort A will consist of 100 CRAC patients with stage II/III resectable disease due for adjuvant chemotherapy.

Cohort B will consist of 30 patients with stage II resectable disease for observation only.

Both cohorts will have a follow up period of up to 2 years, post chemotherapy for cohort A and post resection for cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to give written informed consent
* Histologically or cytologically confirmed CRAC
* Cohort A: colorectal cancer patients with stage II/III resectable disease due for adjuvant chemotherapy OR Cohort B: colorectal cancer patients with stage II resectable disease for observation only
* Age ≥ 18 years
* Treatment with curative intent
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 - 2

Exclusion Criteria:

* Presence of a medical or psychiatric condition, which, in the opinion of the investigator, would potentially pose a risk to the patient when participating in this trial
* Evidence of a metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 CRAC patients with stage II/III resectable disease due for adjuvant chemotherapy.
  30 CRAC patients with stage II resectable disease for observation only.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Disease free survival or progression free survival | Duration of treatment and follow up, expected to be 4 years
  Identify plasma biomarkers with improved sensitivity to predict early recurrence of CRAC and presence of residual occult metastases following completion of adjuvant chemotherapy

SECONDARY OUTCOMES:
Accuracy, sensitivity, specificity and concordance index | Duration of treatment and follow up period, expected to be 4 years
  To validate a panel of predictive and/or prognostic plasma biomarkers, proving its accuracy, sensitivity, specificity and concordance index.
To investigate the correlation between biomarkers identified in plasma samples with the expression of the same biomarkers at tissue level. | For the duration of treatment and follow up, expected to be 4 years
  This allows for further understanding of the role of cancer-related and/or host-related proteins in disease response and progression

CONTACTS AND LOCATIONS:
Locations (14):
- Ireland (14):
  - Beacon Hospital, Bracken Rd, Sandyford Industrial Estate, Dublin 18
  - Our Lady of Lourdes Hospital Drogheda, Drogheda, Louth
  - Bon Secours Hosptial, Cork
  - Cork Universtiy Hospital, Cork
  - Letterkenny General Hospital, Donegal
  - Adelaide & Meath Hospital incorporating National Children's Hoptial (AMNCH), Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St Vincent's Hospital, Dublin
  - Galway University Hospital, Galway
  - Midwestern Regional Hosptial, Limerick, Limerick
  - Sligo General Hospital, Sligo
  - Waterford Regional Hospital, Waterford